CLINICAL TRIAL: NCT06114017
Title: Effect of a Week-long Social Media Abstention on Sustained Attention Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Amber Sousa, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BHS-1894
Record Dates: First submitted 2023-07-24; First posted 2023-11-02 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Attention Difficulties
Keywords: social media; attention; wellbeing

STUDY DESIGN:
Intervention Model Description: Randomized experimental and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Social Media Abstention (Experimental): People in this arm will be encouraged to disable social media and not use social media for one week.
  Interventions: Behavioral: Social Media Abstention
- 2: Control (No Intervention): People in this group will continue their normal behavior in regard to social media use.

INTERVENTIONS:
Behavioral: Social Media Abstention — People will stop or reduce their social media use for one week.
  Arms: 1: Social Media Abstention

SUMMARY:
The current study's goal is to determine if a one-week break from social media in all forms has a beneficial effect on people's attention, as measured by the Sustained Attention to Response Task, executive function as measured by the Stroop test, and well-being.

DETAILED DESCRIPTION:
50 participants between the ages of 18 and 30 years will be recruited for the study via fliers and word of mouth. Following consent procedures, those who choose to participate will be randomized to intervention or control. 25 will be randomly selected to be in the social media group and the other 25 will be selected to go 1 week without engaging with or viewing social media to the best of their ability.

All participants will complete a demographic form at baseline and a survey about their use of social media, as well as the Bergen Social Media Assessment Scale, and the Warwick-Edinburgh Mental Wellbeing Scale. Following that, they will complete the Stroop and the SART, described below. All 50 of them will be asked to take the SART and Stroop (Inquisit Millisecond versions) tests to obtain baseline attention and executive functioning measures. Temporary deletion of social media apps will be supervised by an investigator. Subjects will be given a daily brief report/log to record any use of social media through Redcap. At the end of the week a repeat SART, Stroop, and Warwick-Edinburgh Mental Wellbeing scale will be re-administered. The group that deleted their social media will then be able to redownload their social media if they so choose. A survey about their subjective experience at the conclusion of the week will then be given to all subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* have and regularly use some form of social media
* use on average more than 1 hour of social media a day
* are willing to temporarily delete all social media for 1 week duration

Exclusion Criteria:

* no social media usage
* ADHD or other known conditions that affect attention and/or concentration
* current concussion

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Inquisit Sustained Attention to Response Task (SART) | through study completion, an average of one week
  A 6-minute computerized measure of attention.

SECONDARY OUTCOMES:
Inquisit Stroop Test | through study completion, an average of one week
  A 5-minute measure of executive functions.
Warwick-Edinburgh Mental Wellbeing Scale | through study completion, an average of one week
  A self-report measure of general wellbeing

CONTACTS AND LOCATIONS:
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No